CLINICAL TRIAL: NCT02566564
Title: An Open Label, Single Dose, Dose-escalating Phase I/IIa Study to Determine the Safety and Clinical Effects of Intra-articular Injections of Lopain (MTX-071) in Patients With Chronic Osteoarthritic Knee Joint Pain
Brief Title: Intra-articular Lopain (MTX-071) Phase I/IIa Study in Chronic Osteoarthritic Knee Joint Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MTX-071-P01
Record Dates: First submitted 2015-09-22; First posted 2015-10-02 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open label, single arm (Experimental): Open label, single arm, dose escalating
  Interventions: Drug: Lopain

INTERVENTIONS:
Drug: Lopain — intra-articular injection
  Other Names: MTX-071

SUMMARY:
Phase I/IIa study to determine the safety and clinical effects of intra-articular injections of MTX-071 (Lopain) in patients with chronic osteoarthritic knee-joint pain.

DETAILED DESCRIPTION:
Open label, single-dose, dose-escalating phase I/IIa study to determine the safety and clinical effects of intra-articular injections of MTX-071 (Lopain) in patients with chronic osteoarthritic knee-joint pain.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Written informed consent
* Men or women aged between 40 and 70 years
* At least 40 mm on motion and at least 10 mm at rest on the 100 mm-VAS (Visual Analog Scale) for average arthritic joint pain in the knee to be studied during the last 2 days, with or without pain medication.
* Previously documented radiography showing a Kellgren Lawrence Grade 2 - 4 severity.
* Female patients of childbearing potential or female partners of childbearing potential of male patients must agree to use a reliable contraceptive method for at least one month after the injection of MTX-071.
* Subject is highly likely to comply with the protocol and complete the study.

Exclusion Criteria:

* Knee surgery within 6 months before study start or planned for any time during the next 6 months.
* Any injection into the knee to be studied within the preceding 7 days or trauma to the knee not yet healed.
* History of any clinically significant cardiac, renal, and/or other relevant disease or malignancy.
* History of severe allergic or anaphylactic reactions.
* Pregnancy.
* Major bleeding disorder.
* Clinically significant deviation from the normal laboratory values.
* Clinically significant abnormal ECG
* History of clinically relevant drug/chemical/ substance/alcohol abuse within the past 2 years prior to screening.
* Symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within the past 2 weeks prior to study medication administration.
* Patients positive for human immunodeficiency virus (HIV) antibody, hepatitis C antibody, or for hepatitis B virus surface antigen (HBsAg), tuberculosis.
* Patients who had a corticosteroid injection in the knee to be studied within 3 months prior to baseline or are planned to get a corticosteroid injection within 4 weeks following the injection of MTX-071.
* Vaccination within 60 days prior to study medication administration.
* Systemic immunosuppressant agent within 6 months prior to study medication administration
* Experimental agent within 30 days or ten half-lives, whichever is longer, prior to study medication administration.
* Any other condition, which in the opinion of the investigator, precludes the subject's participation in the trial.
* Patients who are dependent on the sponsor or investigator.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Intensity and severity of AES/SAEs potentially causally related with the study medication | up to 6 months
  overall and per dose level (descriptive statistics) incidence, intensity and severity of AES/SAEs potentially causally related with the study medication

SECONDARY OUTCOMES:
pain relief response: overall and dose response | up to 6 months
  overall and per dose level percentage of patients overall percentage of patients with pain relief response to single intraarticular administration of Lopain (MTX-071) defined as more than a 20% decrease from baseline in mm on the VAS for pain on motion without increase in pain medication
duration of pain relief response: overall and dose response | up to 6 months
  overall and per dose level intra-patients maintenance at 7 days, 1, 3 and 6 months of the pain relief response defined as more than a 20% decrease from baseline in mm on the VAS for pain on motion without increase in pain medication
Acceptance of / satisfaction with treatment as stated by the patients and physicians. (VAS score) | up to 6 months
  per dose level VAS score on acceptance of / satisfaction with treatment as stated by the patients and physicians.
Influence of treatment on functionality of the knee joint and patients' general feeling of health and estimation of daily life conditions (VAS scores) | up to 6 months
  per dose level VAS scores on functionality of the knee joint and patients' general feeling of health and estimation of daily life conditions

CONTACTS AND LOCATIONS:
Overall Officials: Steven Ramael, Principal Investigator — SGS Antwerpen, Belgium
Locations (1):
- SGS Antwerpen, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided